CLINICAL TRIAL: NCT04395560
Title: Highlighting the Benefits of a Screening Protocol Delivered by Orthoptists to Identify Visual Impairment in Children Aged 3 to 4
Acronym: ORTHOPHTALMO
Status: Completed | Type: Observational
Sponsor: Clinique Rive Gauche (Other)
Responsible Party: Sponsor
Other Study IDs: 01/2020; 2020-A00262-37 (Other: ID-RCB)
Record Dates: First submitted 2020-05-13; First posted 2020-05-20 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Visual Impairment in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Visual developmental abnormalities affect 10 to 15% of the population under 6 years of age and leads to amblyopia in 30% of cases if left untreated. Untreated amblyopia in adulthood has consequences on the quality of life of individuals but will also represent a cost to society due to the increased risk of visual impairment.

The screening protocol for this study recommends that a screening examination for amblyopia and amblyogenic factors be routinely performed by an orthoptist in children between 3 and 4 year old. This examination should include, as a minimum, a standardised measurement of visual acuity, a cover test and a measurement of refraction by photoscreener. In the event of a positive screening, the child must then be referred to an ophthalmologist so as to complete an ophthalmological examination.

The aim of this protocol is to propose screening tests usually performed with a high specificity, in order to avoid congestion of ophthalmological services (i.e. by avoiding excessive or unnecessary referral of children to the ophthalmologist) without losing sensitivity by combining several tests.

The orthoptists' role in this screening protocol is to facilitate an extensive screening coverage of the population in this age group, as they are more easily accessed by the patients and more equitably spread in the community than ophthalmologists.

Therefore, by initially screening and then referring less children to the ophthalmologist, the aim is to reduce waiting times in the access of ophthalmological services which could be detrimental in terms of treatment success rates for patients acutely needing care.

Based on the referral of children between 3 and 4 years of age by the orthoptist to an ophthalmologist, the analysis of the data from the standard screening protocol used in our centre will enable us to validate it scientifically. The referral thresholds can thus be secondarily adjusted for each test if the initial objectives are not achieved (specificity > 90% and sensitivity > 87%). The aim of this study is also to observe a change in the patient flow by reducing the volume of consultations with the ophthalmologist currently required based on the present referral rate. The efficiency of the screening protocol by calculating the probable economic gain linked to the modification of the screening circuit will be secondarily studying in this protocol

ELIGIBILITY:
Inclusion Criteria:

* Children from 3 to 4 years old consulting for a screening of visual disorders,
* Patients registered with French social security scheme,
* Not participating in any other clinical study,
* Consent obtained from one of the two parents or the legal representative.

Exclusion Criteria:

* Children whose parent or legal representative is vulnerable according to article L1121-6 of the CSP,
* Children whose parent or legal guardian is under guardianship or trusteeship or under legal protection,
* Children, whose parent or legal guardian is unable to give consent, or is protected by law.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children from 3 to 4 years old, girls or boys, with a medical reason for consultation (paediatric orientation) or parent's request (child's complaint)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-10-04 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
The need to refer the child to an ophthalmologist (YES/NO) | through study completion, an average of 1 year
  the addressing requirements is evaluated by the orthoptist and ophthalmologist based on the patient's chart and clinical examinations

SECONDARY OUTCOMES:
Score of parental satisfaction (algorithmically calculate) | through study completion, an average of 1 year
  Assessed by the Likert scale (satisfaction questionnaire)
The number of ophthalmologic consultations saved | through study completion, an average of 1 year
  Evaluated according to the tariffs of the different nomenclatures of the acts

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Dr Thouvenin, Principal Investigator — Ophtalmologie Rive Gauche
Locations (1):
- Ophtalmologie Rive Gauche, Toulouse, Occitanie, France

REFERENCES:
- [Derived] Lequeux L, Bonifas C, Alby A, Bontron C, Brovelli C, Huygens J, Norbert O, Pey C, Martinez L, Thouvenin Md D. Evaluation of the diagnostic parameters of the amblyopia and risk factors for amblyopia screening protocol in 3-year-olds according to recommendations from the French Association for Pediatric Ophthalmology and Strabismus (AFSOP) compared with reference ophthalmological examination: the ORTHOPHTALMO study. Strabismus. 2025 Jun;33(2):93-103. doi: 10.1080/09273972.2024.2422418. Epub 2024 Nov 6. PMID 39506219